CLINICAL TRIAL: NCT04322253
Title: Investigation of the Pharmacokinetics, Safety, and Tolerability of Neladenoson Bialanate in Subjects With Hepatic Impairment (Classified as Child Pugh A and B) and in Age-, Weight-, and Gender-matched Healthy Subjects, Following a Single Oral Dose in a Single-center, Non-randomized, Non-controlled, Non-blinded Study
Brief Title: Study on the Safety of Neladenoson Bialanate, How it is Tolerated and the Way the Body Absorbs, Distributes and Gets Rid of the Study Dug Given as a Single Oral Dose in Participants With Liver Impairment and Healthy Participants Matched for Age-, Gender-, and Weight
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The cessation of the development project for neladenoson bialanate.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15139; 2017-000482-74 (EudraCT Number)
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Pharmacology, Clinical
MeSH Terms: interventions — neladenoson bialanate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neladenoson bialanate, mild hepatic impairment (Experimental): Subjects with Child Pugh score 5 or 6 received a single immediate-release (IR) tablet dose of 10 mg neladenoson bialanate in the fasted state
  Interventions: Drug: Neladenoson bialanate (BAY 1067197)
- Neladenoson bialanate, moderate hepatic impairment (Experimental): Subjects with Child Pugh score 7-9 received a single IR tablet dose of 10 mg neladenoson bialanate in the fasted state
  Interventions: Drug: Neladenoson bialanate (BAY 1067197)
- Neladenoson bialanate, control group (Experimental): Healthy subjects matched for age, gender and body weight received a single IR tablet dose of 10 mg neladenoson bialanate in the fasted state
  Interventions: Drug: Neladenoson bialanate (BAY 1067197)

INTERVENTIONS:
Drug: Neladenoson bialanate (BAY 1067197) — 10 mg as a single IR tablet dose. Active metabolite: BAY 84-3174

SUMMARY:
Neladenoson bialanate is currently under clinical development for a condition in which the heart has trouble pumping blood through the body (chronic heart failure). Liver impairment is a condition in which the liver is not working as well as they should. The goal of the study is to learn more about the safety of neladenoson bialanate, how it is tolerated and the way the body absorbs, distributes and excretes the study dug given as a single oral dose neladenoson bialanate in participants with liver impairment and healthy participants matched for age-, gender-, and weight

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Male and female Caucasian subjects between 18 and 79 years of age (both inclusive) with a body mass index above/equal 18.0 and below/equal 34.0 kg/m² Subjects with hepatic impairment
* Subjects with documented liver cirrhosis confirmed by histopathology, e.g., previous liver biopsy, laparoscopy, ultrasound, or fibroscan
* Subjects with hepatic impairment as per Child Pugh system
* Subjects with stable liver disease during the last 2 months Healthy subjects
* Healthy subjects with mean age and body weight not varying by more than ±10 years and ±10 kg from the groups of subjects with mild and moderate hepatic impairment, respectively.

Exclusion Criteria:

* Medical history of continent ileostomy.
* Febrile illness within 1 week prior to admission to study center.
* Known hypersensitivity to the study drug (active substances or excipients of the preparation).
* Subjects with diagnosed malignancy within the past 5 years.
* Use of any systemic or topical medicine or substances which oppose the study objectives or which might influence them, in particular:

Starting from screening on, but minimum from 2 weeks before the study drug administration until the follow-up visit:

* CYP3A4 inducers
* CYP3A4 inhibitors
* Potent CYP2C8 inhibitors
* Major uridine diphosphate-glucuronosyltransferase isoenzyme 1A1 (UGT1A1) substrate (irinotecan)

On the day of administration of neladenoson bialanate:

* Major breast cancer resistance protein (BCRP) substrates
* Regular daily consumption of more than 500 mL of usual beer or the equivalent quantity of of more than 2 units of alcohol in another form - Intake of ethanol containing food and beverages from 48 h prior to admission to the study center until 96 h after study drug administration, afterwards not more than 2 units of alcohol per day until follow-up examination.
* Intake of food and beverages containing grapefruit or pomelo from 14 days prior to study drug administration up to the last time point of PK sampling.
* Therapies (e.g. physiotherapy, acupuncture, etc.) within 1 week before study drug administration.
* Positive urine drug screening.
* Positive results for human immune deficiency - Abnormal (clinically significant) thyroid stimulating hormone (TSH).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
fu for BAY 84-3174 | At 4 hours after study drug administration
  Fraction of free (unbound) drug in plasma or serum after single dose administration
AUC for BAY 84-3174 | Pre-dose up to 49 days after study drug administration
  Area under the concentration vs. time curve from zero to infinity after single dose administration
AUCu for BAY 84-3174 | Pre-dose up to 49 days after study drug administration
  AUC of unbound drug after single dose administration
AUCnorm for BAY 84-3174 | Pre-dose up to 49 days after study drug administration
  AUC divided by dose per body weight after single dose administration
Cmax for BAY 84-3174 | Pre-dose up to 49 days after study drug administration
  Maximum observed drug concentration in measured matrix after single dose administration
Cmax,u for BAY 84-3174 | Pre-dose up to 49 days after study drug administration
  Cmax of unbound drug after single dose administration
Cmax,norm for BAY 84-3174 | Pre-dose up to 49 days after study drug administration
  Cmax divided by dose per body weight after single dose administration

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) | Up to 49 days after study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/